CLINICAL TRIAL: NCT07152704
Title: Clitoral Sensitivity Enhancement With Hyperstacking of Er:YAG SMOOTH Mode
Brief Title: Clitoral Sensitivity Enhancement With Laser
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Espacio Gaspar Clinic (Other)
Responsible Party: Principal Investigator, Adrian Gaspar, Principal Investigator, Espacio Gaspar Clinic
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CLIT / 01
Record Dates: First submitted 2025-08-26; First posted 2025-09-03 (Actual); Last update posted 2025-09-11 (Actual); Status verified 2025-08

CONDITIONS: Decreased Clitoral Sensitivity
Keywords: non-ablative; Er:YAG laser; clitoral atrophy; hyperstacking; sexual health; orgasm; clitoris
MeSH Terms: conditions — Orgasm

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Active therapy with non-ablative Er:YAG laser (Experimental): Patients underwent three laser sessions with non-ablative SMOOTH Er:YAG laser, with 20 days interval between sessions
  Interventions: Device: Active therapy with non-ablative Er:YAG laser

INTERVENTIONS:
Device: Active therapy with non-ablative Er:YAG laser — three intravaginal and vulvar/clitoral treatments within 60 days

SUMMARY:
The purpose of this clinical trial is to evaluate whether non-ablative Er:YAG laser treatment can improve decreased clitoral sensitivity in adult women who report this concern. Effectiveness and safety will be assessed after each laser session and again at a 2-month follow-up visit.

DETAILED DESCRIPTION:
This study is designed to investigate whether non-ablative Er:YAG laser treatment can improve clitoral sensitivity in adult women who report decreased sensitivity. Reduced clitoral sensitivity can negatively impact sexual response, orgasm, and quality of life, yet effective treatment options are limited.

The primary goal of this clinical trial is to determine the effectiveness and safety of non-ablative Er:YAG laser treatment for women experiencing decreased clitoral sensitivity. Specifically, the study aims to assess:

The degree to which laser treatment enhances vaginal and clitoral sexual response, the time required to achieve noticeable improvements in sexual response, the impact of treatment on orgasmic function and patient satisfaction with the treatment process and outcomes.

Participants will undergo three laser treatment sessions, with evaluations conducted at a 2-month follow-up. Both effectiveness (improvements in sexual response and satisfaction) and safety outcomes will be carefully monitored.

By exploring this minimally-invasive therapeutic option, the study seeks to provide new insights into the management of decreased clitoral sensitivity and to help identify safe and effective approaches for improving sexual health in women.

ELIGIBILITY:
Inclusion Criteria:

* above 18 years
* sexually active at least once per month

Exclusion Criteria:

* anorgasmia
* pregnancy
* urinary tract infections
* genital infectious diseases of other etiology (HPV, molluscum contagiosum, syphilis, HIV, etc.)
* genital bleeding
* collagenopathies
* ongoing chemotherapy
* active genital cancer
* patients undergoing pelvic radiotherapy
* any genital or extragenital pathology that may interfere with treatment
* patients who have limitations in performing a follow-up to this study
* patients with psychiatric disorders that may be difficult to treat
* patients who have a contraindication to vaginal laser treatments

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 133 (Actual)
Dates: Start 2022-03-01 (Actual); Primary Completion 2022-12-31 (Actual); Study Completion 2022-12-31 (Actual)

PRIMARY OUTCOMES:
Change of bothersome symptoms (decreased intensity of clitoral/vaginal response, decreased time of good sexual response, decreased orgasm sensation) | Change from Baseline at 2 months after last intervention
  Evaluation of clitoral sensitivity change was performed 2 months after the last treatment session. Patients answered a five-point Likert scale (from 0 to 4) questionnaire.

SECONDARY OUTCOMES:
Patient satisfaction with 5-point Likert scale | Each visit included recording of any adverse effect. Patients were instructed to report and adverse effect that may have occured during the whole duration of the study.
  Patients were asked to assess their global satisfaction with the treatment on a 5-point Likert scale (1-Very unsatisfied, 2-Unsatisfied, 3-Neutral, 4-Satisfied, 5-Very satisfied).
Recording of frequency and severity of adverse effects related to laser treatment | From Baseline to 2 months after last intervention
  Each visit included recording of any adverse effect. Patients were instructed to report and adverse effect that may have occured during the whole duration of the study.

CONTACTS AND LOCATIONS:
Overall Officials: Adrian Gaspar, MD, Principal Investigator — Espacio Gaspar Clinic
Locations (1):
- Uroclinica, Mendoza, Argentina

IPD SHARING:
Plan to Share IPD: No